CLINICAL TRIAL: NCT02034435
Title: Endogenous Renin-Angiotensin-Aldosterone System and Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, James Matt Luther, M.D., MSCI, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 131139
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Sodium-Restricted; Salts; Eplerenone; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (4):
- Aim1-Low Sodium then High Sodium (Active Comparator): Subjects will be provided with a low sodium diet from the Vanderbilt Clinical Research Center that will be controlled for salt content.
  Participants will be given low sodium diet (50mEq/d) and Placebo tablets for 8 days and assessments will be made, washout and then cross over to a low sodium diet (50mEq/d) plus Salt tables (150mEq) for 8days and assessments will be made.
  Interventions: Other: Low Salt diet plus Placebo tablet; Other: Low Sodium diet plus Salt tablet
- Aim 1-high salt diet then low salt diet (Active Comparator): Subjects will be provided with a diet from the Vanderbilt Clinical Research Center that will be controlled for salt content.
  Participants will be given low sodium diet (50mEq/d) and Salt tables (150mEq) for 8 days and assessments will be made, washout and then cross over to a low sodium diet (50mEq/d) plus Placebo tablets for 8days and assessments will be made.
  Interventions: Other: Low Salt diet plus Placebo tablet; Other: Low Sodium diet plus Salt tablet
- Aim2- low salt diet and epleronone then amlodipine (Active Comparator): Subjects on a low salt diet will receive Epleronone 50mg for 8 days and assessments will be made, then cross over to a low salt diet with Amlodipine 5mg for 8days and assessments will be made.
  Interventions: Other: Low Salt diet plus Placebo tablet; Drug: Epleronone; Drug: Amlodipine
- aim2- low salt diet and amlodipine then epleronone (Active Comparator): Subjects on a low salt diet will receive Amlodipine 5mg for 8 days and assessments will be made, then cross over to a low salt diet with Epleronone 50mg for 8days and assessments will be made.
  Interventions: Other: Low Salt diet plus Placebo tablet; Drug: Epleronone; Drug: Amlodipine

INTERVENTIONS:
Other: Low Salt diet plus Placebo tablet
Other: Low Sodium diet plus Salt tablet
  Arms: Aim 1-high salt diet then low salt diet; Aim1-Low Sodium then High Sodium
Drug: Epleronone — 50mg daily
  Other Names: Inspra
  Arms: Aim2- low salt diet and epleronone then amlodipine; aim2- low salt diet and amlodipine then epleronone
Drug: Amlodipine — 5mg daily
  Other Names: Norvasc
  Arms: Aim2- low salt diet and epleronone then amlodipine; aim2- low salt diet and amlodipine then epleronone

SUMMARY:
Aim 1.Test the hypothesis that activation of the endogenous renin-angiotensin-aldosterone system impairs glycemic control via effects on insulin sensitivity and insulin secretion.

Aim 2. Test the hypothesis that activation of the endogenous renin-angiotensin-aldosterone system impairs insulin secretion and insulin sensitivity via an mineralocorticoid-receptor dependent mechanism.

DETAILED DESCRIPTION:
In aim 1 subjects are randomized to cross over between an 8 day high salt and 8 day low salt diet and assessments are made.

In aim 2, subjects are randomized to a 2x2 cross over study with an 8 day low salt diet and either eplerenone 50mg or amlodipine 5mg.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects, 18 to 70 years of age, inclusive
2. For female subjects, the following conditions must be met:

   1. postmenopausal status for at least 1 year, or
   2. status-post surgical sterilization, or
   3. if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing prior to drug treatment and on every study day.
3. Metabolic Syndrome as defined by the presence of > 3 of the following:

   1. Systolic Blood Pressure > 130 mm Hg OR Diastolic Blood Pressure > 85 mm Hg.
   2. Glucose Intolerance (Fasting Plasma Glucose ≥ 100 mg/dL)
   3. Increased triglyceride level > 150mg/dL (1.7mmol/L)
   4. Decreased levels of HDL cholesterol (For males, less than 40 mg/dL; For females, less than 50 mg/dL)
   5. Waist circumference (For males, greater than 40 inches; For females, greater than 35 inches)

Exclusion Criteria:

1. type 1 Diabetes
2. Type II Diabetes
3. Impaired renal function
4. Prior allergies to medications used in the study protocol
5. Screening plasma potassium >5.5 mmol/L or sodium <135 mmol/L
6. Cardiovascular disease
7. Use of hormone replacement therapy
8. Breast-feeding
9. Treatment with anticoagulants
10. History of serious neurologic disease
11. History or presence of immunological or hematological disorders
12. Diagnosis of asthma requiring use of inhaled beta agonist
13. Clinically significant gastrointestinal impairment
14. Impaired hepatic function
15. Hematocrit <35%
16. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal antiinflammatory drugs
17. Treatment with chronic systemic glucocorticoid therapy
18. Treatment with lithium salts
19. History of alcohol or drug abuse
20. Treatment with any investigational drug in the 1 month preceding
21. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
22. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Luther, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim1-Low Sodium Then High Sodium: Subjects will be provided with a low sodium diet from the Vanderbilt Clinical Research Center that will be controlled for salt content.
  Participants will be given low sodium diet (50mEq/d) and Placebo tablets for 8 days and assessments will be made, washout and then cross over to a low sodium diet (50mEq/d) plus Salt tables (150mEq) for 8days and assessments will be made.
  Low Salt diet plus Placebo tablet
  Low Sodium diet plus Salt tablet
- Aim 1-High Sodium Then Low Sodium: Subjects will be provided with a diet from the Vanderbilt Clinical Research Center that will be controlled for salt content.
  Participants will be given low sodium diet (50mEq/d) and Salt tables (150mEq) for 8 days and assessments will be made, washout and then cross over to a low sodium diet (50mEq/d) plus Placebo tablets for 8days and assessments will be made.
  Low Salt diet plus Placebo tablet
  Low Sodium diet plus Salt tablet
- Aim2- Low Sodium Diet and Epleronone Then Amlodipine: Subjects on a low salt diet will receive Epleronone 50mg for 8 days and assessments will be made, then cross over to a low salt diet with Amlodipine 5mg for 8days and assessments will be made.
  Low Salt diet plus Placebo tablet
  Epleronone: 50mg daily
  Amlodipine: 5mg daily
- Aim2- Low Sodium Diet and Amlodipine Then Epleronone: Subjects on a low salt diet will receive Amlodipine 5mg for 8 days and assessments will be made, then cross over to a low salt diet with Epleronone 50mg for 8days and assessments will be made.
  Low Salt diet plus Placebo tablet
  Epleronone: 50mg daily
  Amlodipine: 5mg daily
Period: Overall Study
Arm/Group | Aim1-Low Sodium Then High Sodium | Aim 1-High Sodium Then Low Sodium | Aim2- Low Sodium Diet and Epleronone Then Amlodipine | Aim2- Low Sodium Diet and Amlodipine Then Epleronone
Started | 13 | 15 | 7 | 9
Aim 1 | 13 | 15 | 0 | 0
Aim 2 | 0 | 0 | 7 | 9
Completed | 11 | 13 | 7 | 8
Not Completed | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Illness | 0 | 2 | 0 | 0
Not completed — Inadequate IV access | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aim 1: Low Sodium and High Sodium diet crossover
- Aim 2: Eplerenone and Amlodipine crossover
- Total: Total of all reporting groups
Arm/Group | Aim 1 | Aim 2 | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [29 to 56] | 46 [43 to 56] | 45 [40 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 16 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 24 | 15 | 39
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: Hyperglycemic clamp- acute insulin response (AIR) during time 0-10 minutes
Time Frame: After 8 days of diet or drug
Population: Participants with metabolic syndrome
Measure: Median (Inter-Quartile Range); unit: uU/mL*10min
Groups:
- Aim 1- Low Sodium: Low Sodium diet (50mEq/d)
- Aim 1- High Sodium: Low sodium diet (50mEq/d) plus sodium tablet (150 mEq/d)
- Aim 2- Eplerenone: Low sodium diet (50mEq/d) plus Eplerenone
- Aim 2- Amlodipine: Low sodium diet (50mEq/d) plus Amlodipine
Arm/Group | Aim 1- Low Sodium | Aim 1- High Sodium | Aim 2- Eplerenone | Aim 2- Amlodipine
Number analyzed (Participants) | 28 | 28 | 15 | 16
uU/mL*10min | 293.1 [186.9 to 369.4] | 234.7 [161.3 to 479.7] | 330.8 [268.2 to 481.5] | 300.4 [177.8 to 477.8]

2. Primary Outcome: Insulin Sensitivity
Description: Hyperinsulinemic clamp- glucose infusion rate during insulin administration
Time Frame: after 8 days of diet or medication
Population: Participants with metabolic syndrome
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Aim 1- Low Sodium | Aim 1- High Sodium | Aim 2- Eplerenone | Aim 2- Amlodipine
Number analyzed (Participants) | 28 | 28 | 15 | 16
mg/kg/min | 6.6 [5.5 to 7.6] | 6.9 [6.1 to 7.6] | 6.4 [5.8 to 8.2] | 6.3 [5.4 to 7.7]

ADVERSE EVENTS:
Time Frame: Monitoring during 1 week of intervention/drug, washout period, and during cross-over to 1 week of remaining intervention/drug. Monitoring for adverse events continued up to 2 weeks after study completion.
Arm/Group | Aim 1- Low Sodium | Aim 1- High Sodium | Aim 2- Eplerenone | Aim 2- Amlodipine
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/28 | 10/28 | 3/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aim 1- Low Sodium (N=28) | Aim 1- High Sodium (N=28) | Aim 2- Eplerenone (N=16) | Aim 2- Amlodipine (N=16)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) — Headache during study
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) — Nausea
viral illness (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Unrelated viral or other illness
Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness/Lightheadedness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Low glucose (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — low glucose after clamp, resolved
IV infiltration or malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — bruising, swelling, or pain at IV site
numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — temporary numbess in hand, resolved spontaneously
discomfort with swallowing pill (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — temporary discomfort when swallowing tablets
Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — rectal fissure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02034435/Prot_SAP_000.pdf